CLINICAL TRIAL: NCT06063408
Title: The Effectiveness of Cognitive Functional Therapy in Adults With Chronic Neck Pain: A Pragmatic Randomized Controlled Trial
Brief Title: The Effectiveness of Cognitive Functional Therapy in Adults With Chronic Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European University Cyprus (Other)
Responsible Party: Principal Investigator, George Ploutarchou, Principal Investigator, European University Cyprus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0101100333
Record Dates: First submitted 2023-09-05; First posted 2023-10-02 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Chronic Pain
Keywords: Chronic neck pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Functional Therapy (Experimental): Participants will received in this group four main component:
  1. Pain education, cognitive education, explanation about their health condition, self management education
  2. Graded exposure to painful movements or activities
  3. Movement therapy targeted to their functional integration
  4. Lifestyle programme.
  Interventions: Behavioral: Cognitive Functional Therapy
- Conventional Therapy (Active Comparator): Participants will received in this group four main component:
  1. Tens therapy
  2. Massage to cervical and shoulder area
  3. Relaxation techniques
  4. Posture exercises
  5. Workplace education
  Interventions: Behavioral: Conventional Therapy

INTERVENTIONS:
Behavioral: Cognitive Functional Therapy — Cognitive functional therapy (CFT) is a novel intergraded behavioral approach for individualizing the management of spinal pain, targeting the bio-psycho-social factors of rehabilitation, and enabling the patient to self-manage the condition.
  CFT lies within the broad spectrum of the biopsychosocial approach for the management of spinal pain. CFT uses a multidimensional clinical reasoning framework with aim to enable the clinician to identify modifiable components of the condition, evaluate patients' behavioral responses to pain, and compose and drive a tailored rehabilitation program mainly based on self-management. The intervention is comprised by the interplay on "making sense of pain", "exposure with control", and "lifestyle change".
  Other Names: CFT
  Arms: Cognitive Functional Therapy
Behavioral: Conventional Therapy — Each individual session involve a combination of pain management with electrotherapy, massage and relaxation techniques. Also include some posture exercise these will be targeted on body alignment to the neutral position, and strengthening the whole neck area. strengthening program will be include isometrics on all cervical movements with a band which progressively increase the resistance of the band by change it and process to exercise against the band resistant. The relaxation/mindfulness component will take place at the end of each class and will involve breathing and relaxation of the body.
  Other Names: CT
  Arms: Conventional Therapy

SUMMARY:
The aim of this study was to compare the effectiveness of Cognitive Functional Therapy compared with Conventional Therapy in treating adults with chronic neck pain

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informer consent will undergo 1 week screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility criteria will be randomized in a single- blind manner (assessor), in a 1:1 ration to cognitive functional therapy or conventional therapy twice a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* Pain in neck area for more than 3 months
* Pain in NPRS more than 40/100
* Independently mobile (with or without aids), to be capable of participating in a rehabilitation program twice a week

Exclusion Criteria:

* Serious psychological pathology
* recently surgery on shoulder or neck area (<6 months)
* Pain relieving procedures such as injection based therapy (e.g epidurals) and day case procedures (e.g rhizotomy) in the last 3 months
* Pregnancy
* Rheumatologic/inflammatory disease (e.g. rheumatoid arthritis (RA), ankylosing spondylitis (AS), psoriatic arthritis, lupus, scheuermann's disease)
* Progressive neurological disease (e.g. multiple sclerosis (MS), parkinson's disease (PD), motor neuron disease (MND)
* Unstable cardiac conditions
* Red flag disorders like malignancy/cancer, acute traumas like fracture (<6 months ago) or infection, spinal cord compression/cauda equina

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale | Baseline (after randomization), at 4th week (after 8th session), at 8th week (after 16th session), 3 months (after randomization)
  Measured pain intensity with 0 no pain and 100 the worst pain ever.
Neck Disability Index | Baseline (after randomization), at 4th week (after 8th session), at 8th week (after 16th session), 3 months (after randomization)
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life.
  0= no disability 100= severe disability

SECONDARY OUTCOMES:
Fear Avoidance Beliefs Questionnaire | Baseline (after randomization), at 4th week (after 8th session), at 8th week (after 16th session), 3 months (after randomization)
  The Fear-Avoidance Beliefs Questionnaire (FABQ) is a patient reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability.
  The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96. A higher score indicates more strongly held fear avoidance beliefs.
Short Fort 12 | Baseline (after randomization), at 4th week (after 8th session), at 8th week (after 16th session), 3 months (after randomization)
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
EurQqol 5 | Baseline (after randomization), at 4th week (after 8th session), at 8th week (after 16th session), 3 months (after randomization)
  An EQ-5D health state is the set of responses to the 5 dimensions of EQ-5D, as completed by a patient or respondent.
  Values are anchored at 1 (full health) and 0 (a state as bad as being dead) as required by their use in economic evaluation. Values less than 0 represent health states regarded as worse than a state that is as bad as being dead.
Range of motion | Baseline (after randomization), at 4th week (after 8th session), at 8th week (after 16th session), 3 months (after randomization)
  Range of motion in all cervical movement, flexion, extension, side flexion, rotations
Isometric Strength | Baseline (after randomization), at 4th week (after 8th session), at 8th week (after 16th session), 3 months (after randomization)
  Strength in all cervical movement, flexion, extension, side flexion, rotations

CONTACTS AND LOCATIONS:
Locations (1):
- European University of Cyprus, Nicosia, Engomi, Cyprus